CLINICAL TRIAL: NCT06232434
Title: An Open Prospective Randomized Clinical Study of the Effectiveness, Tolerability and Safety of a Single Intraperitoneal Use of the Drug "Prospidelong, Powder for the Preparation of a Gel for Topical Use, 1000 mg in Vials, Package No. 1" in Patients With Disseminated Gastric Cancer, Phase I-II
Acronym: ИНТЕЛОН-02
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Research Institute for Physical Chemical Problems of the Belarusian State University (Other)
Collaborators: N.N. Alexandrov National Cancer Centre (Other Government); Unitary Enterprise UNITEHPROM BSU (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ИНТЕЛОН-02
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer With Peritoneal Dissemination
Keywords: gastric cancer with peritoneal dissemination; prospidin; dextran phosphate
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): after diagnostic laparotomy/laparoscopy, a single intraperitoneal administration of the study drug Prospidelong, produced by UNITEHPROM BSU, Republic of Belarus, further in accordance with the protocols of the Ministry of Health of the Republic of Belarus for the treatment of patients with the corresponding pathology, systemic chemotherapy in accordance with the clinical protocol "Diagnosis and treatment of malignant neoplasms" (approved by Resolution of the Ministry of Health of the Republic of Belarus No. 60 of 07/06/2018).
  Interventions: Drug: Prospidelong; Procedure: chemotherapy
- Comparison group (Placebo Comparator): after diagnostic laparotomy/laparoscopy, systemic chemotherapy in accordance with the clinical protocol "Algorithms for the diagnosis and treatment of malignant neoplasms" (approved by Resolution of the Ministry of Health of the Republic of Belarus No. 60 of 07/06/2018), namely the section regulating the treatment of patients suffering from metastatic gastric cancer with the degree of prevalence of the tumor process corresponding to sT1-4N0-3M1.
  Interventions: Procedure: chemotherapy

INTERVENTIONS:
Drug: Prospidelong — Prospidium chloride (in the form of prospidelong (a mixture of prospidium chloride and dextran sodium salt phosphate containing carbamate groups in a 1:1 ratio)) - 1000 mg.
  Arms: Experimental arm
Procedure: chemotherapy — after diagnostic laparotomy/laparoscopy, systemic chemotherapy in accordance with the clinical protocol "Algorithms for the diagnosis and treatment of malignant neoplasms" (approved by Resolution of the Ministry of Health of the Republic of Belarus No. 60 of 07/06/2018), namely the section regulating the treatment of patients suffering from metastatic gastric cancer with a degree of prevalence tumor process corresponding to sT1-4N0-3M1

SUMMARY:
It is planned to conduct an open-label, prospective, randomized clinical study of the efficacy, tolerability and safety of a single intraperitoneal administration of the investigational drug Prospidelong at a dose of 4000 mg (2000 mg in terms of prospidium chloride) in patients with disseminated gastric cancer.

In total, the study plans to include 120 patients aged 18 to 75 years inclusive, including 60 patients in the study group and 60 in the comparison group. The study consists of daily examination of patients throughout the entire period of hospitalization and subsequent visits.

DETAILED DESCRIPTION:
It is planned to conduct an open-label, prospective, randomized clinical study of the efficacy, tolerability and safety of a single intraperitoneal administration of the investigational drug Prospidelong at a dose of 4000 mg (2000 mg in terms of prospidium chloride) in patients with disseminated gastric cancer.

In total, the study plans to include 120 patients aged 18 to 75 years inclusive, including 60 patients in the study group and 60 in the comparison group. The study consists of daily examination of patients throughout the entire period of hospitalization and subsequent visits.

Inclusion - preliminary interview with the patient and signing of informed consent.

Informed consent is the free and voluntary expression of the subject's desire to participate in a specific study after receiving information about all aspects of this study that are significant for the subject's decision to participate, and in the case of minors and incapacitated subjects, the permission or consent of their legal representatives to include such subjects into the study. Informed consent is documented by signing and dating the informed consent form.

Signed and dated informed consent must be obtained from each patient or, if the patient is unable to make an informed decision due to health reasons, from the patient's spouse/close relative (close relatives include parents, adult children, siblings, grandparents) , grandchildren), and the patient's signed informed consent to participate in the study must additionally be obtained as soon as his health condition allows it.

Before signing informed consent, all potential participants should be informed of the nature and purpose of the study, including possible risks and unwanted effects, and given sufficient time to read and understand the information presented. The researcher should answer any questions that arise. The researcher must also sign an informed consent form. After signing, one copy of the informed consent is given to the patient (the patient's spouse/close relative) and one copy remains at the center for storage in the Researcher's file.

Preparatory period - includes screening patients for compliance with inclusion and exclusion criteria, determining the initial condition of the patient. During screening, a medical history will be taken and the patient's date of birth, age and gender will be recorded. When collecting anamnesis, you should clarify data on concomitant diseases and medications used to treat the main and concomitant diseases, drug intolerance, and allergic reactions.

During screening, the patient's medications and procedures performed over the past 30 days must also be recorded. Registration of concomitant therapy for the main and concomitant diseases is carried out at each visit. All changes in the treatment regimen for the underlying disease (changes in the standard therapy received by the patient as part of rehabilitation treatment in the postoperative period and during systemic chemotherapy drug treatment after discharge from the hospital) and in the treatment of concomitant diseases are recorded: changes in the dose and frequency of administration of previously prescribed drugs, prescription new drugs.

After signing the informed consent and screening, patients undergo a general clinical examination in accordance with the clinical protocol "Algorithms for the diagnosis and treatment of malignant neoplasms" (approved by Resolution of the Ministry of Health of the Republic of Belarus No. 60 of 07/06/2018).

The scope of research before treatment includes:

* Fibrogastroscopy with tumor biopsy and morphological examination of the biopsy material (if necessary, x-ray examination of the stomach) - for no more than 30 days before inclusion.
* ECG.
* Ultrasound examination (ultrasound) of the abdominal organs - for no more than 30 days before inclusion.
* X-ray examination of the lungs - within no more than 60 days before inclusion.
* Computer tomography of the chest and abdominal cavity (within no more than 60 days before inclusion). If this study is available, performing an ultrasound of the abdominal organs and an X-ray examination of the lungs is not mandatory.
* Palpation of peripheral lymph nodes, digital examination of the rectum - for no more than 7 days before inclusion.
* Examination by a gynecologist for women - no later than 6 months before inclusion.
* Laboratory tests: blood group, Rh factor, seroreaction to syphilis, general blood test (hemoglobin, erythrocytes, leukocytes, segmented neutrophils, platelets), general urinalysis, biochemical blood test (protein, creatinine, urea, bilirubin, AST, ALT), coagulogram (activated partial thromboplastin time, thrombin time, fibrinogen) - for no more than 7 days before inclusion.

According to indications: fibrocolonoscopy, laparoscopy, irrigoscopy, angiography, MRI, scintigraphy of skeletal bones, computed tomography - for no more than 7 days before inclusion.

Preliminary selection. Based on the results of the preoperative examination, a preliminary selection of patients with resectable gastric cancer is carried out.

The final selection is carried out intraoperatively based on the results of the abdominal cavity revision (see above). Patients with the presence of peritoneal dissemination, confirmed by morphological examination, are selected. The scope of surgical intervention will be limited to biopsy of areas of the peritoneum with disseminates. Randomization of patients will be carried out by an employee of the department of automated control systems of the Republican Scientific and Practical Center for OMR named after. N.N. Aleksandrova using the "Randomization" software based on random number generation. The result of randomization will be confirmed by protocols of the established form. During randomization, patients will be divided into the following groups: main (experimental) and control group. Patients of the main group, after placing a control drainage in the abdominal cavity, will undergo intraperitoneal application of the study drug Prospidelong at a dose of 4000 mg. Patients in the control group did not undergo intraperitoneal administration of Prospidelong.

Individual registration cards (IRCs) are created for patients included in a clinical trial.

Recruitment of patients into the groups will be done using a sequential enrollment method. Patients excluded from the study for any reason will not be replaced.

Treatment period Intraperitoneal use of the study drug Prospidelong will be a single dose. Subsequent treatment of patients will be carried out in accordance with the clinical protocol "Algorithms for the diagnosis and treatment of malignant neoplasms" (approved by Resolution of the Ministry of Health of the Republic of Belarus No. 60 of 07/06/2018).

The scope of research in the study groups in the postoperative period will include:

* survey and physical examination of the patient (includes analysis of the patient's general condition, objective status, determination of body temperature and heart rate, identification of symptoms of irritation and inflammation of the peritoneum) - daily during the entire period of the patient's stay in the hospital;
* detailed general blood test (hemoglobin, erythrocytes, leukocytes, segmented neutrophils, platelets) for 1.5±1, 10±2, 90±7, 180±7, 270±7, 360±7, 540±7, 720± 7 days after surgery;
* biochemical blood test (total protein, creatinine, urea, bilirubin, AST, ALT) for 1.5±1, 10±2, 90±7, 180±7, 270±7, 360±7, 540±7, 720 ±7 days after surgery;
* general urine analysis 1 day, 10±2, 90±7, 180±7, 270±7, 360±7, 540±7, 720±7 days after surgery;
* Ultrasound (or CT if necessary) of the abdominal organs 90±7, 180±7, 270±7, 360±7, 540±7, 720±7 days after surgery;
* ECOG score 1.5±1, 10±2, 90±7, 180±7, 270±7, 360±7, 540±7, 720±7 days after surgery.

Deviations in the timing of ultrasound and CT of the abdominal cavity are allowed if progression of the tumor process is suspected (CT is performed only if progression of the disease is suspected and other research methods are not informative).

After using the study drug Prospidelong, the researcher evaluates the immediate and immediate results and enters the evaluation data into the CRF. The assessment of the necessary parameters is carried out in the hospital after surgery, as well as during subsequent visits to the patient for a follow-up examination within the specified time frame.

At each study visit, the patient's complaints will be assessed by the study physician.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer without transition to the esophagus with peritoneal dissemination sT1-4N0-3M1.
* Life expectancy of at least 6 months
* Physical status on the ECOG scale 0 - 1.
* The age of patients is from 18 to 75 years.
* Absence of severe concomitant diseases in the decompensation stage.
* Availability of written informed consent from the patient to participate in the study.
* The ability of the patient and the personnel caring for him to comply with the instructions of the research physician and comply with the study design.

Exclusion Criteria:

* Pregnancy and lactation.
* The presence of a primary multiple (synchronous or metachronous) malignant tumor. The exception is for patients who were treated for basal cell or squamous cell skin cancer, cervical cancer in situ, or other tumors more than 5 years ago and are expected to be completely cured.
* Presence of severe concomitant diseases in the stage of decompensation;
* Family relationships between the patient and the center staff.
* Allergy to components of the study drug.
* Refusal of the patient from the proposed treatment method.
* Presence of heart disease class III or IV according to the New York Heart Association classification or a history of myocardial infarction within 6 months before the 1st day of the study.
* Any history of epileptic seizures.
* Severe diseases, including those with severe symptoms, untreated inflammatory and infectious processes, due to which the patient cannot receive treatment in accordance with the study protocol.
* Chronic liver and/or kidney failure.
* Legal incapacity or other circumstances due to which the patient or his immediate family are unable to understand the nature, scope and possible consequences of the treatment being carried out
* Socioeconomic or geographic circumstances that cannot guarantee adequate compliance with protocol requirements for treatment and follow-up.
* History of abuse of alcohol or any chemical substances for 2 years up to the 10th day before the start of the study.
* Patient participation in another clinical trial.

Non-inclusion criteria based on survey data:

* Acute bleeding from the tumor.
* Level of peripheral blood leukocytes less than 1.5 × 109 per l, platelets less than 75.0 × 109 per l.
* Hemoglobin less than 80g per l.
* Positive tests for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Severe liver dysfunction - AST and ALT levels exceed the upper limit of normal by 5 times or more, bilirubin greater than or equal to 2.0 mg per dL (34.2 µmol per L).
* Severe renal impairment - creatinine clearance less than 30 ml per minute, calculated using the Cockcroft-Gault formula - or the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula.
* Diabetes mellitus in a state of clinical and metabolic decompensation.

Criteria for exclusion (dropout) from the study:

* Individual intolerance to drugs included in the treatment regimen.
* The patient's desire to stop participating in the study.
* Serious adverse events occurring in the patient during the study.
* Violation by the patient of the research conditions of the investigational medicinal product (non-compliance).
* Pregnancy.
* Detection of a second malignant tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
increased survival | through study completion, an average of 2 years
  The criterion for the effectiveness of a single intraperitoneal administration of the investigational drug Prospidelong in patients with disseminated gastric cancer will be an increase in progression-free survival after use of the investigational drug Prospidelong. Progression of disseminated peritoneal tumors with documented evidence of an increase in the grade of disseminated peritoneal tumors (compared to baseline) on non-invasive intrascopic imaging (CT or MRI) will be considered as events in the calculation of progression-free survival for this clinical trial. abdominal cavity) and/or second-look laparotomy. In the latter case, assessment of the peritoneal tumor index P.H. will be mandatory. Sugarbaker. Second-look laparotomy will be planned in patients with no evidence of progression of the tumor process according to multislice computed tomography or magnetic resonance imaging of the abdominal cavity.

SECONDARY OUTCOMES:
Ultrasound and/or computed tomography of the abdominal cavity (if necessary) | through study completion, an average of 2 years
  the progression or stabilization of the disease is assessed during treatment (systemic chemotherapy) by identifying distant metastases (liver, lungs) or an increase in their number, the appearance or increase in the amount of ascitic fluid in the dynamics of observation and/or the presence of disseminates
detailed general blood test | through study completion, an average of 2 years
  Blood samples will be collected for the analysis of hemoglobin, erythrocytes, leukocytes, segmented neutrophils, platelets level
blood chemistry | through study completion, an average of 2 years
  Blood samples will be collected for the analysis of total protein, creatinine, urea, bilirubin, AST, ALT level

CONTACTS AND LOCATIONS:
Locations (1):
- The state institution N. N. Alexandrov National Cancer Centre of Belarus, Minsk, Minsk City, Belarus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solomevich SO, Bychkovsky PM, Yurkshtovich TL, Golub NV, Mirchuk PY, Revtovich MY, Shmak AI. Biodegradable pH-sensitive prospidine-loaded dextran phosphate based hydrogels for local tumor therapy. Carbohydr Polym. 2019 Dec 15;226:115308. doi: 10.1016/j.carbpol.2019.115308. Epub 2019 Sep 9. PMID 31582057